CLINICAL TRIAL: NCT06976814
Title: Facial Palsy Treatment: Investigating the Most Effective Modality of Therapy for Recovery?
Brief Title: Facial Palsy Treatment
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Mohammed Sajid Hussain, Director of Rehabilitation, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-20-1167
Record Dates: First submitted 2025-04-15; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Facial Palsy; Stroke Rehabilitation
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neuro muscular electrical stimulation arm (Experimental)
  Interventions: Other: Neuro muscular electrical stimulation
- Beckmann Oral Motor Exercise Arm (Experimental)
  Interventions: Other: Beckmann's oral motor exercises
- Neuro Muscular Electrical Stimulation Arm + Beckmann Oral Motor Exercise Arm (Experimental)
  Interventions: Other: Neuro muscular electrical stimulation; Other: Beckmann's oral motor exercises

INTERVENTIONS:
Other: Neuro muscular electrical stimulation — electrical stimulation to facial nerve to improve facial palsy
  Arms: Neuro Muscular Electrical Stimulation Arm + Beckmann Oral Motor Exercise Arm; Neuro muscular electrical stimulation arm
Other: Beckmann's oral motor exercises — Oral motor exercises to improve facial palsy.
  Arms: Beckmann Oral Motor Exercise Arm; Neuro Muscular Electrical Stimulation Arm + Beckmann Oral Motor Exercise Arm

SUMMARY:
The Primary objective of the study is to investigate the most effective treatment modalities available to speech language pathologist as well as movement difference by comparing them.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1st stroke
* Hemorrhagic stroke
* Ischemic stroke
* Right hemispheric stroke
* Left hemispheric stroke
* Normal cognitive skills (Based on Montreal cognitive assessment MOCA)
* Normal Language (Not Aphasic)
* Normal swallowing

Exclusion Criteria:

* Patients with Bell's palsy
* Facial trauma
* Post otitis media surgeries
* Neoplasm, malignant or tumor cell invasion of facial nerve
* Cognitive impairment
* Patients with aphasia
* Patients on defibrillator cardiac devices
* Patients with pacemakers or any other type of cardiac devices
* Multiple strokes

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Sunnybrook Facial Grading System | Patients were enrolled for 30sessions as per the protocol. Participants were given 5 sessions in a week. Patients were assessed as baseline upon enrollment into the study and re-assessed beginning of each week.
  Upon enrollment Sunnybrook is given as baseline. The minimum score a patient may score is 20 out of 100. The higher the score the better (means patient has minor facial asymmetry). Each participant/patient was planned for 30sessions. Baseline score was recorded and beginning of each week Sunnybrook was given and new score was recorded by the same clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar, Qatar

IPD SHARING:
Plan to Share IPD: No
Patient privacy